CLINICAL TRIAL: NCT02602301
Title: The Effect of Intravenous Oxytocin Infusion Using Different Diluents on Neonatal Bilirubin & Sodium Levels .A Prospective Randomized Controlled Trial.
Brief Title: The Effect of Intravenous Oxytocin Infusion Using Different Diluents on Neonatal Bilirubin & Sodium Levels
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed El-Sharkawy, kasr el ainy hospital,kasr el ainy street ,cairo egypt, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: oxytocin
Record Dates: First submitted 2015-11-08; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: oxytocin
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): group A that included 109 women in whom labour was augmented by IV infusion of oxytocin using isotonic saline 0.9%,
  Interventions: Drug: Oxytocin
- 2 (Active Comparator): group B that included 109 women in whom labour was augmented by IV infusion of oxytocin using glucose 5% .
  Interventions: Drug: Oxytocin
- 3 (Placebo Comparator): Group C in which 109 women continued their labour course without any further augmentation.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — different oxytocin diluents and effect on fetal bilirubin&sodium levels.
  Other Names: syntocinon

SUMMARY:
Objective: To evaluate the relationship between intravenous (IV) infusion of oxytocin using either saline 0.9% or glucose 5% & neonatal Bilirubin & sodium level.

Study Design: A randomized case - controlled study. Setting: The Obstetrics and Gynecology casuality department of Kasr El Aini hospital (Cairo University - Egypt)

DETAILED DESCRIPTION:
This prospective randomized case-controlled study was performed at the Obstetrics and Gynecology causality Department of Kasr El Aini University hospital, Cairo University, Egypt in the period from November 2015 to March 2016. The study was approved by the Hospital Ethical Committee. Informed consents were obtained from all patients after explanation of the aim of the study & the potential risks. The study was not supported by any pharmacological company.

327 multigravidas with singleton living healthy fetus presented to the casuality department with spontaneous onset of labour & gave birth through the vaginal route were enrolled in the study. They were randomized into 3 groups: group A that included 109 women in whom labour was augmented by IV infusion of oxytocin using isotonic saline 0.9%, group B that included 109 women in whom labour was augmented by IV infusion of oxytocin using glucose 5% & group C (control group) in which 109 women continued their labour course without any further augmentation.

Inclusion criteria included: maternal age between 20 & 35 years old, gestational age 37 to 40 weeks (confirmed by a reliable date for the last menstrual period and 1st trimester ultrasound scan), vertex presentation of the fetus & intact membranes. Women who had chronic or pregnancy induced diseases or any contraindication to vaginal delivery (e.g. malpresentation, contracted pelvis & placenta previa) were excluded. Additional exclusion criteria included rhesus (Rh) negative or (O) blood group mothers, prolonged labour (> 12h), fetal distress, instrumental delivery (forceps or vacuum extraction), abnormal fetal growth (IUGR or macrosomia), non-reassuring initial fetal CTG & epidural analgesia. Neonates with one or more of the following criteria were excluded: Apgar score < 5 or <7 at one minute or five minutes respectively, low birth weight (< 2.5 kg), birth trauma or abnormal G6PD enzyme levels.

For all patients, full history was taken followed by complete physical examination & obstetric ultrasound. Initial baseline CTG was done to confirm fetal wellbeing. Patient was then randomized to one of the three groups. 5 units oxytocin was placed in 500 cc of isotonic saline 0.9% or 5% glucose With the beginning of active phase (defined as fully effaced cervix with 3-4 cm dilatation), the investigator gave the patient either 5 units oxytocin placed in 500 cc of isotonic saline 0.9% (group A) or 5% glucose (group B). The rate of infusion in both groups was 2.5 mIU/min of oxytocin intravenous drip with the dose increased by 2.5 mIU/ml every 20min till effective uterine contractions establishment (defined as the presence of 3 forceful uterine contractions over 10 mins span). Amniotomy was done at cervical dilatation ≥ 6 cm if spontaneous rupture of membranes did not occur. Opioid analgesia was given after the amniotomy (meperidine hydrochloride 50 mg IM). Oral fluid intake was not restricted in all patients.

Participants were monitored in bed together with fetal wellbeing surveillance using continuous CTG monitoring. A partogram was maintained throughout labour and vaginal examinations were conducted and recorded every 2 hours.

Following fetal delivery, cord was clamped within 2 minutes from birth Sodium and initial bilirubin levels were measured in the cord. Umbilical cord blood samples (10 ml) were obtained from the placental site of divided umbilical cord into heparin test tubes and plasma was separated immediately. Sodium, initial haemtocrit & bilirubin levels were measured. All babies were breastfed. Neonatal capillary blood (obtained by heel prick) bilirubin and haemtocrit concentrations were remeasured on day 1 and 2. Sodium measurement was done using flame photometry while bilirubin level was determined using spectrophotometry.

Data collected included total volume of fluid & total oxytocin dose administered till delivery, neonatal Apgar score at birth (1 & 5 minutes), birth weight, cord sodium, haemtocrit & bilirubin levels at birth and neonatal plasma haemtocrit & bilirubin levels on day 1 & 2.

ELIGIBILITY:
Inclusion Criteria:

* maternal age between 20 & 35 years old, gestational age 37 to 40 weeks (confirmed by a reliable date for the last menstrual period and 1st trimester ultrasound scan), vertex presentation of the fetus & intact membranes

Exclusion Criteria:

* Women who had chronic or pregnancy induced diseases or any contraindication to vaginal delivery (e.g. malpresentation, contracted pelvis & placenta previa) were excluded. Additional exclusion criteria included rhesus (Rh) negative or (O) blood group mothers, prolonged labour (> 12h), fetal distress, instrumental delivery (forceps or vacuum extraction), abnormal fetal growth (IUGR or macrosomia), non-reassuring initial fetal CTG

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 327 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
neonatal bilirubin level | 5 months.
  11/2015 to March 2016

SECONDARY OUTCOMES:
neonatal APGAR score | 5 months
  11/2015 to 3 /2015

CONTACTS AND LOCATIONS:
Overall Officials: Kasr El Ainy, Study Director — kasr el ainy street,cairo,egypt; mohamed el sharkawy, M.D., Principal Investigator — 72 A Manial street,4thfloor.